CLINICAL TRIAL: NCT03390907
Title: Hybrid APC Assisted EMR for Large Colon Polyps to Reduce Local Recurrence : A Prospective Data Collection Study
Brief Title: Hybrid APC Assisted EMR for Large Colon Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, John M. Levenick, Assistant Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008877
Record Dates: First submitted 2017-12-29; First posted 2018-01-04 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Colon Polyp; Colon Adenoma; Colon Cancer
Keywords: Colon polyp; EMR; Hybrid-APC; Laterally spreading tumor
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a pilot study design in which patients with non-pedunculated large polyps ≥ 20mm undergoing EMR will be recruited. Following standard EMR all patients will undergo adjuvant Hybrid Argon Plasma Coagulation (APC) of the base edges of the polypectomy site to fulgurate any potential microscopic residual disease.
Masking Description: Following Standard EMR all patients will undergo adjuvant Hybrid Argon Plasma Coagulation (APC) of the base and edges of the polypectomy site to fulgurate any potential microscopic residual disease.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hybrid APC (Experimental): Hybrid APC ( Erbe Hybrid APC) design for ablation of abnormal tissue in GI tract.
  Interventions: Device: Hybrid APC

INTERVENTIONS:
Device: Hybrid APC — Following standard EMR Hybrid Argon Plasma Coagulation (APC) of the base and edges of the polypectomy site to fulgurate any potential microscopic residual disease.

SUMMARY:
The purpose of this study to evaluate and examine whether use of Hybrid Argon Plasma Coagulation (APC) as an adjunct to endoscopic mucosal resection (EMR) will reduce the risk of residual or recurrent neoplasia at 6 months. Hybrid APC is an existing FDA approved device used to assist with ablation of abnormal tissue anywhere in the GI tract.

DETAILED DESCRIPTION:
Colon Cancer is a major disease that effects more than 1 million people per year globally. Adenomatous polyps have been identified as the main precursor leading to colorectal cancer. Colon cancer screening is the best way to detect and remove large, often asymptomatic polyps. Early detection and resection of these colorectal polyps can prevent the development of colon cancer. Endoscopic mucosal resection (EMR) is a technique used for resection of medium to large colon polyps. In this technique, fluid is injected into the submucosa creating a cushion between the mucosa and the muscularis propria. An electrocautery snare is then deployed to resect the polyp in a single (en-bloc) or multiple (piecemeal) pieces. Most polyps >2 cm are resected in piecemeal way. Although EMR is now considered standard of care with a successful resection rate of 85 % and low risk of complication (3-10% bleeding and 1% perforation), this technique has inherent deficiencies, especially piecemeal EMR. Recurrence rates following piecemeal EMR can be as high as 20%. Resection of scarred polyps using this technique is particularly challenging due to the non-lifting of the polyp. Endoscopic submucosal dissection (ESD) is an alternative approach that aims to remove non- pedunculated precancerous or cancerous lesions over 20 mm in one piece (en-bloc resection rate of 89.95% and lesion recurrence rate of 0.7%). However, due to its technical complexity and high complication risk (mainly bleeding and perforation, with complication rates approximately 8%), it is not the current standard of care and only performed by experts in the technique.

Hybrid Argon plasma coagulation (APC) is a new technique in which the endoscopist reinjects the submucosa with fluid to create a cushion (normal saline/ diluted adrenaline and /or sodium hyaluronate solution) to protect the muscle layer and then ablation is done using spray argon coagulation to treat any microscopic residual disease that is the seed for local recurrence. Previous studies have shown that this technique is a safe and easily applicable technique to complete resection for recurrent polyps after first EMR.

Investigators hypothesize that with Hybrid APC assisted EMR there will be a decrease in recurrence rate after 6 months and it will be more effective compared to the standard EMR procedure.

This is a pilot study in which patients with non-pedunculated large polyps ≥ 20mm undergoing endoscopic mucosal resection (EMR) will be recruited. Following standard EMR all patients will undergo adjuvant Hybrid Argon Plasma Coagulation (APC) of the base and edges of the polypectomy site to fulgurate any potential microscopic residual disease. Resected polyps will be sent to the pathology laboratory where pathologist determine the final diagnosis of the polyps as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged ≥18 and ≤89 of any gender, ethnicity and race referred to endoscopy for resection of large colon polyps
* Patients with a ≥20mm colon non-pedunculated polyp
* Ability to give written informed consent

Exclusion Criteria:

* Patients with known (biopsy proven) invasive carcinoma in a potential study polyp
* Pedunculated polyps (as defined by Paris Classification type Ip or Isp)
* Patients with ulcerated depressed lesions (as defined by Paris Classification type III)
* Patients with inflammatory bowel disease
* Patients who are receiving an emergency colonoscopy
* Poor general health (ASA class>3)
* Patients with coagulopathy with an elevated INR ≥1.5, or platelets <50
* Poor bowel preparation
* Target sign or perforation during initial EMR
* Need for ESD for complete resection prior to APC
* Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Levenick, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in Hershey Medical Center with a known ≥ 20mm polyp detected at a prior colonoscopy who were referred for colonoscopy procedure were identified as potential study participants.
Period: Overall Study
Arm/Group | Hybrid APC
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participant population was 10% (n=4) African American and 90% (n=36) with 100% (n=40) non-Hispanic/Latino population
Arm/Group | Hybrid APC
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Measurement of polyps in mm [Mean (Standard Deviation); unit: mm] — Included polyps were a median size of 27 mm (IQR: 14.5 mm) and predominantly located in the ascending colon (31.8%), cecum (25.0%), and transverse colon (20.5%).
  mm | 35.2 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Having Complete Resection
Description: The primary outcome of interest will be the percentage of participants having complete resection at 6 months.
Time Frame: 6 months post initial procedure
Measure: Count of Participants; unit: Participants
Groups:
- Hybrid APC: Hybrid APC ( Erbe Hybrid APC) design for ablation of abnormal tissue in GI tract.
  Hybrid APC: Following standard EMR Hybrid Argon Plasma Coagulation (APC) of the base and edges of the polypectomy site to fulgurate any potential microscopic residual disease.
  0% of recurrence in 32 cases who completed post-procedure colonoscopy 6 month follow-up.
Arm/Group | Hybrid APC
Number analyzed (Participants) | 40
Participants | 40

2. Secondary Outcome: Measure of Within 30 Days of Procedure Adverse Events ( Post-polypectomy Bleeding and Post-polypectomy Syndrome)
Description: The secondary outcome of interest will be measure of major adverse event rate, mainly post-polypectomy bleeding and post-polypectomy syndrome
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Hybrid APC
Number analyzed (Participants) | 40
Participants | 3

ADVERSE EVENTS:
Time Frame: At 30 days following the initial resection, the research coordinator called each patient to assess for any signs of post-procedural adverse events.
Arm/Group | Hybrid APC
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 3/40
Other Adverse Events (participants affected / at risk) | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hybrid APC (N=40)
Bleeding (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03390907/Prot_SAP_000.pdf